CLINICAL TRIAL: NCT01046435
Title: Effects of Periodontal Therapy on Markers of Systemic Inflammation in Subjects at Cardiovascular Disease Risk
Brief Title: Effects of Periodontal Therapy on Systemic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Nestor J. Lopez, University of Chile Faculty of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FONDECYT 1061070
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2006-05

CONDITIONS: Periodontal Disease; Cardiovascular Disease; Type 2 Diabetes; Obesity; Metabolic Syndrome
Keywords: periodontitis; cardiovascular disease; diabetes
MeSH Terms: conditions — Periodontal Diseases; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome; Periodontitis; Diabetes Mellitus | interventions — Metronidazole; Amoxicillin; Periodontal Index

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supragingival scaling plus placebo (Placebo Comparator): Plaque control instructions, supra gingival scaling and two placebos
  Interventions: Procedure: metronidazole and amoxicillin; Procedure: Two placebos
- Root planing plus antibiotics (Experimental): Plaque control instructions, subgingival scaling,root planing, metronidazole 250 mg and amoxicillin 500 mg. three times a day for 7 days
  Interventions: Procedure: metronidazole and amoxicillin; Procedure: Two placebos

INTERVENTIONS:
Procedure: metronidazole and amoxicillin — Metronidazole 250 mg three times a day per 7 days
  Other Names: Non-surgical periodontal therapy
Procedure: Two placebos — Two placebos 3 times a day for 7 days
  Other Names: Community periodontal treatment

SUMMARY:
The purpose of this study is to determine if treating periodontal infections (gum disease) will reduce markers of systemic inflammation in patients at risk of cardiovascular diseases.

DETAILED DESCRIPTION:
Aims: To determine the effects of periodontal treatment on systemic markers of inflammation in subjects with risk of coronary heart disease.

Methods: The current study is a randomized, double blind clinical trial, with two treatment groups.

Eligible participants will be allocated by restricted randomization using the minimization method to the treatment group or to the control group. The treatment group will receive periodontal therapy consisting of instructions of plaque control, supra and subgingival scaling and root planing, oral systemic metronidazole (250 mg) plus amoxicillin (500 mg) tid for 7 days. The control group will receive plaque control instructions, supragingival scaling and two placebos. The study plan to enroll 160 participants, 80 in ech arm, over a 6-month period. Follow-up clinic visits will be scheduled to occur every 3 months after finishing treatment. Baseline and follow-up clinic visits will include periodontal examination, blood collection and medical and dental histories. The following biochemical markers will be determined at baseline and at 3, 6, 9 and 12 months posttherapy: total, LDL and HDL lipoprotein cholesterol and triglycerides, glycemia, high sensitivity C-reactive protein, fibrinogen, erythrocyte sedimentation rate and white blood cells count. In diabetic patients, glycosylated hemoglobin will be also assessed.

The study will be conducted in a public health center in Santiago, Chile. To be eligible for the study, participants have to be older than 35 years and fulfill the medical and periodontal criteria. For the medical criteria participants have to have dyslipidemia, and at least one of the following coronary heart disease risk factors: obesity, smoking, diabetes, hypertension.

The periodontal inclusion criteria are: no history of periodontal treatment, the presence of at least 14 natural teeth, with at least 4 teeth with interproximal sites with probing depth equal or higher than 4 mm and concomitant attachment loss equal or higher than 3 mm, and >30 % of sites with bleeding on probing.

The outcomes measures will be levels of serum C-reactive protein, fibrinogen, erythrosedimentation rate, white blood cell count.The outcomes will be measured at 0, 3,6,9, and 6 months after periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosis of marginal periodontitis
* No history of periodontal treatment
* At least 14 natural teeth present
* Dyslipidemia
* And at least one of the following factors:

  * obesity
  * diabetes
  * smoking, hypertension

Exclusion Criteria:

* Rheumatoid arthritis
* Any type of cancer in the previous 2 years
* Pregnancy and lactation
* Indication of the use of antibiotic for invasive procedures
* Use of antibiotics in previous three months.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Serum levels of C-reactive protein, fibrinogen,erythrosedimentation rate and white blood cell count | 0, 3, 6, 9 and 12 months after therapy

SECONDARY OUTCOMES:
Clinical periodontal parameters: probing depth, bleeding on probing, clinical attachment level | 0, 3, 6, 9 and 12 months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nestor J. Lopez, DDS, Principal Investigator — University of Chile; Antonio Quintero, DDS, Principal Investigator — University of Chile; Carola Ibieta, DDS, Study Chair — University of Chile; Carlos Y Valenzuela, DMS, PhD, Study Chair — University of Chile; Lilian Jara, MsB, PhD, Study Chair — University of Chile; Marcelo Llancaqueo, DMS, Study Chair — University of Chile
Locations (1):
- Dra Eloisa Díaz Health Center, Metropolitan Northen Health Service, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- See also: Related Info — http://www.fondecyt.cl/578/channel.html